CLINICAL TRIAL: NCT05639634
Title: The Efficacy of Chlorella Supplementation on Health and Performance Following a 12-week Training Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21745/002
Record Dates: First submitted 2022-10-24; First posted 2022-12-06 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Sedentary; Overweight
MeSH Terms: conditions — Sedentary Behavior; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chlorella Supplementation and Exercise (Experimental): Supplementation with Chlorella (1.5 g/d) with a physical exercise program for 12 weeks
  Interventions: Dietary Supplement: Chlorella supplementation; Other: 12 week cardiovascular training programme
- Chlorella Supplementation (Experimental): Supplementation with Chlorella (1.5 g/d) only for 12 weeks. No exercise programme
  Interventions: Dietary Supplement: Chlorella supplementation
- Placebo Supplementation and Exercise (Placebo Comparator): Supplementation with Placebo - microcrystalline cellulose (1.5 g/d) with a physical exercise program for 12 weeks
  Interventions: Other: 12 week cardiovascular training programme; Dietary Supplement: Placebo Supplementation
- Placebo Supplementation (Placebo Comparator): Supplementation with Placebo - microcrystalline cellulose (1.5 g/d) only for 12 weeks. No exercise programme
  Interventions: Dietary Supplement: Placebo Supplementation

INTERVENTIONS:
Dietary Supplement: Chlorella supplementation — Supplementation with Chlorella (1.5 g/d) in 3 capsules for 12 weeks.
  Arms: Chlorella Supplementation; Chlorella Supplementation and Exercise
Other: 12 week cardiovascular training programme — Participants will be asked to complete a 12 week cycling training programme. This will consist of 4 X 50 min sessions per week. Each exercise session will include a warm-up phase (~ 5 min), a main physical conditioning phase (~ 40 min), and a cool-down phase (~ 5 min).
  Arms: Chlorella Supplementation and Exercise; Placebo Supplementation and Exercise
Dietary Supplement: Placebo Supplementation — Supplementation with Placebo - microcrystalline cellulose (1.5 g/d) in 3 capsules for 12 weeks.
  Arms: Placebo Supplementation; Placebo Supplementation and Exercise

SUMMARY:
Algae are an emerging functional food source that are gaining traction and popularity in biopharmaceutical, nutraceutical, and biotechnology industries. They are a diverse and complex species that comprise an abundant breadth of micronutrients (multiple vitamins, minerals, fatty acids, and amino acids) that can possibly promote human health. One such popular algae is chlorella, a unicellular dark green organism, which can be readily bought in health stores worldwide. Although there is some promising data to suggest chlorella supplementation can alleviate cardiovascular risk factors and improve VO2max from supplementation alone, an area which has particularly limited existing literature is the possible ergogenic and health influence of chlorella supplementation combined with a controlled training programme in sedentary and overweight populations. Given that such populations are susceptible to increased risk of developing associated diseases (cardiovascular disease, diabetes, hypertension) and possess poor diets, there is a need to investigate the possible synergistic effect of a training programme and supplementation of algae further. Furthermore, there is growing evidence to suggest that supplementation with algae may have a beneficial effect on cognitive function, primarily owed to antioxidant and anti-inflammatory mechanisms. Therefore, the purpose of this study aims to assess the efficacy of chlorella supplementation on VO2max, blood lipid profiles, cognitive function and body composition following a 12-week training programme. Briefly, in a double blind, randomised, placebo-controlled trial, participants will be randomly allocated into 1 of 4 groups (A. Exercise + Chlorella, B. Exercise + Placebo, C. Control + Chlorella, D. Control + Placebo).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50
* Classified a sedentary (<30 minutes of moderate intensity exercise for <3 days per week for 3 months) and/or overweight (BMI = 25 +)
* Be willing to complete a 12-week training programme

Exclusion Criteria:

* Individuals taking blood thinners.
* Known allergies to algae/mould and iodine.
* Taking immunosuppressant medication
* Regularly ingesting algae
* Smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Changes in cardiovascular fitness (VO2max) | At baseline, week 6 and at week 12
  Changes in cardiovascular fitness variables as measured by a Cardio Pulmonary Exercise Test.
Changes in blood lipid profiling | At baseline, week 6 and at week 12
  Assessing changes in blood lipids (Triglycerides, cholesterol, low-density lipoprotein, High-density lipoprotein)

SECONDARY OUTCOMES:
Changes in cognitive function (simple reaction time) | At baseline, week 6 and at week 12 (before and after exercise)
  Assessing changes in simple reaction time (m/s & number of errors) using the Gorilla Experiment Builder on a laptop.
Changes in cognitive function (inhibition) | At baseline, week 6 and at week 12 (before and after exercise)
  Assessing changes in inhibition (m/s & number of errors) using the Gorilla Experiment Builder on a laptop.
Changes in cognitive function (endogenous and exogenous attending) | At baseline, week 6 and at week 12 (before and after exercise)
  Assessing changes in endogenous and exogenous attending (m/s & number of errors) using the Gorilla Experiment Builder on a laptop.
Changes in cognitive function (context memory) | At baseline, week 6 and at week 12 (before and after exercise)
  Assessing changes in source and context memory (m/s & number of errors) using the Gorilla Experiment Builder on a laptop. spatial anticipation
Changes in cognitive function (spatial anticipation) | At baseline, week 6 and at week 12 (before and after exercise)
  Assessing changes in spatial anticipation (m/s & number of errors) using the Gorilla Experiment Builder on a laptop.
Changes in body composition variables | At baseline, week 6 and at week 12
  Assessing changes in body composition variables using the Tanita. Weight (kg) and height (cm) will be combined to report BMI in kg/m^2.
Changes in body composition variables (fat & lean mass percentage) | At baseline, week 6 and at week 12
  Assessing changes in body fat mass (Body Fat mass %) and lean mass in percentage (Lean mass %) using the Tanita.
Changes in body composition variables (fat free and muscle mass) | At baseline, week 6 and at week 12
  Assessing changes in fat free mass (kg) and muscle mass (kg) using the Tanita.
Changes in blood pressure | At baseline, week 6 and at week 12
  Assessing changes in blood pressure (mmHg). Systolic and diastolic, using the ABP-Monitor Mobil-O-Graph NG
Changes in pulse wave velocity | At baseline, week 6 and at week 12
  Assessing changes in pulse wave velocity (PWV) using the ABP-Monitor Mobil-O-Graph NG.
Changes in total vascular resistance | At baseline, week 6 and at week 12
  Assessing changes in total vascular resistance (TVR) using the ABP-Monitor Mobil-O-Graph NG.
Changes in augmentation index | At baseline, week 6 and at week 12
  Assessing changes in augmentation index (Alx) using the ABP-Monitor Mobil-O-Graph NG.
Changes in augmentation pressure | At baseline, week 6 and at week 12
  Assessing changes in augmentation pressure using the ABP-Monitor Mobil-O-Graph NG.
Changes in lactate | At baseline, week 6 and at week 12
  Assessing changes in lactate at rest, peak, +5mins post, +10mins post, +30mins post
Changes in biomarkers for brain health | At baseline, week 6 and at week 12
  Assessing changes in Brain-Derived Neurotrophic Factor (before exercise at rest and 30-mins post peak exercise)
Changes in Nitrate/Nitrite | At baseline, week 6 and at week 12
  Assessing changes in plasma Nitrate and Nitrite concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Tom Gurney, Principal Investigator — University College, London
Locations (1):
- University Colllege London (ISEH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No